CLINICAL TRIAL: NCT00193752
Title: Para-Aortic Lymph Nodal Staging and Evaluation of Treatment Outcome by 18F-fluorodeoxyglucose Positron Emission Tomography (FDG-PET) in Advanced Cervical Cancer
Brief Title: Para-Aortic Lymph Nodal Staging & Evaluation of Treatment Outcome by 18F FDG-PET in Advanced Cancer Cervix
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Umesh Mahantshetty, Professor, Radiation Oncology, Tata Memorial Hospital
Other Study IDs: TMH/205/2004/Cx_PET STUDY
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Cancer of Cervix
Keywords: FDG-PET Imaging; Cervical Cancer; Post-treatment evaluation; Para-aortic Nodal Staging; Extended field Radiation; Extended field IMRT
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: PET IMAGING — PET imaging in cervical cancers to predict, prognosticate outcome in cervical cancers

SUMMARY:
18F-fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Imaging has been extensively used in the evaluation of various malignancies and is rapidly being recognized as a mandatory investigations. 18F-fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Imaging has also been tried in cervical cancers with excellent results for detection of both pelvic and extra-pelvic disease in terms of sensitivity and specificity. Till date, PET Imaging has been reported to have highest sensitivity and specificity for detection of disease and treatment failures compared to other non-invasive investigations available. Treatment decisions (Localized RT Vs Extended RT) will be according to the results of PET Scans. The treatment response, outcome and follow-up will be labelled according to the PET Scan results and will be directed for treatment accordingly.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Carcinoma Cervix is the commonest malignancy and a leading cause of cancer mortality seen in Indian women. At Tata Memorial Hospital, Carcinoma Cervix constitutes approximately 10% of all cancers (1). Nearly 85% of the patients present with advanced stages (FIGO Stage II/III). The main stay of treatment has traditionally been radical radiation therapy with 80-90% of patients requiring radiation in their lifetime and over decades the survival rates have achieved a plateau of 30 - 55% at 5 years. In patients with advanced stages (stages IIB to IVA), 15 - 38% have para-aortic lymph nodal metastases (2). Identification of para-aortic nodal status allows modification of radiation therapy fields to include this nodal disease, which, because of intestinal morbidity, is not routinely included in the treatment field by most of the Radiation Oncologists. Extended field radiation therapy that includes the para-aortic nodes is associated with a 31% to 50% 5 year-survival, depending on the location and extent of para-aortic nodal metastasis and the likelihood of controlling the pelvic disease (3-5) Therefore, in advanced cervical cancer, it has been reported that progression-free survival is significantly related to para-aortic lymph node metastasis (6-8). In a collective series of Gynecologic Oncology Group protocols, Para aortic nodal status was the most significant indication of recurrence (6).

A number of noninvasive modalities have been used to evaluate the status of para-aortic nodal metastasis. The introduction of Computed Tomographic (CT) Scanning in the mid-1970s provided a method of para-aortic nodal disease evaluation (9). CT Scanning has been widely used for clinical staging, but its sensitivity for nodal metastasis is only 44% (10). In contrast to CT, which primarily relies on the morphologic criteria, FDG-PET can non-invasively assess metabolic activity in cancers and metastatic lesions. The differentiation capability for malignant lesions of FDG-PET is not compromised by using morphologic size criteria. Even malignant lesions less than 1 cm in diameter that manifest high FDG uptake can be differentiated from nonmalignant tissue by using PET. Therefore, FDG-PET can detect metastatic para-aortic lymph nodes in patients with advanced cervical cancer whose lymph nodes have not been abnormally enlarged.

Many published data have previously reported the clinical value of 18F FDG PET for imaging the primary tumor, staging the nodal and visceral involvement, and also detecting a recurrent disease (11-19). Rose et al. (11) used FDG-PET for evaluating nodal metastasis in locally advanced cervical cancer before surgical staging, with a sensitivity of 75% and a specificity of 92% to detect the metastases of para-aortic lymph nodes. They found that the accuracy of FDG-PET was greater than that of CT in detecting the para-aortic lymph nodal metastasis. In a similar series, Wu et al. have reported a sensitivity of 85.7%, a specificity of 94.4%, and an accuracy of 92% with FDG PET to detect para-aortic lymph nodal metastasis in patients with advanced cervical cancer and negative abdominal CT findings. Grigsby et al. (12) demonstrated that FDG-PET detects more abnormal lymph node regions than does CT, and that FDG-PET findings are a better predictor of survival than those of CT in patients with cervical cancer.

Magnetic Resonance Imaging (MRI) has also been reviewed in evaluating both the primary disease at cervix and also para-aortic nodal staging. MRI has been recognized as an important imaging modality for the management of cervical cancer because of its multiplanar capability, distinct tissue contrast characteristics using various pulse sequences, and excellent tissue contrast, particularly between tumor and surrounding normal tissues. However, PET findings were most often compared to CT results, while MRI is nowadays considered as the modality of choice for staging the primary tumor (20,21). Only one study by Narayan et al. has compared the respective value of MRI and PET for staging loco-regionally advanced cervical cancer (22). Their study found that the primary tumor was similarly detected by the two imaging techniques with a sensitivity of 100%. On the other hand, except for small-volume metastases, PET had a sufficiently high positive predictive value (91%) in the pelvis and para-aortic region, to obviate lymph node sampling. More recent studies have shown that the 3D quantitative imaging-based method of tumor size assessment using MRI is highly accurate in determining actual tumor size and extent (23-27) and may be superior to clinical palpation in predicting local tumor control (23,25,28) Conversely, MRI accuracy was insufficient for nodal management. If MRI remains the modality of choice for evaluating the loco-regional status of the primary tumor, metabolic imaging i.e FDG PET seems particularly useful for staging, in one session, extra pelvic nodal metastases. Thus, PET may have a significant impact on treatment decision-making.

Identification of para-aortic nodal status allows modification of radiation therapy fields to include this nodal disease. Stehman et al. previously demonstrated the prognostic importance of para-aortic nodal status in locally advanced cervical carcinoma (6). In advanced cervical cancer, it has been reported that progression-free survival is significantly related to para-aortic lymph node metastasis (6-8). Recent studies have shown a survival benefit in patients with positive para-aortic nodes treated by extended-field irradiation and concurrent radio-sensitizing chemotherapy (29-31).

PET is also of great value for optimally confirming a complete remission and detecting a recurrence non-invasively in post-treatment follow-up. More recently, positron emission tomography (PET) with the glucose analogue, 18 F-fluorodeoxyglucose (FDG) has demonstrated promising results in evaluating tumor response and predicting survival after primary treatment with radiation therapy or chemotherapy for several tumor types, including head-and-neck cancer, breast cancer, seminoma, colorectal cancer, lymphoma, and lung cancer (33-40). Recently, Grigsby et al have reported the role of FDG PET in posttherapy surveillance monitoring in a series of 75 patients with cervical cancer. They have concluded that FDG-PET is a valuable tool to evaluate the response of both at primary and its lymph node disease after radiation therapy and chemotherapy and for the Post-Rx surveillance of patients to detect asymptomatic recurrence (41).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous carcinoma or adenocarcinoma of cervix
* Performance index WHO grade 0 or 1
* Patients below 65 years of age
* FIGO Stage IIB / IIIB
* Normal ECG and Cardiovascular system
* Normal hematological parameters
* Normal renal and liver function tests
* Normal Blood Sugar levels / Controlled Diabetes

Exclusion Criteria:

* Co-morbid conditions like medical renal disease
* Past History of Phobia for MRI Examination
* Medical or Psychological condition that would preclude Investigations / Treatment
* H/o Previous treatment / Pregnancy
* Patient unreliable for treatment completion and follow-up Investigations.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hisotologically proven cervical cancers with FIGO II-IIIB eligible for the study will be invited for the study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2015-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
PET Scan for Para-Aortic Staging in Carcinoma Cervix | 5 years
Clinical (FIGO), MRI, and PET - Abdomen and Pelvis Correlation | 5 years
Volumetric Correlation of Local Disease by PET and MRI | 5 years
Radiotherapy Response Evaluation and Post therapy Surveillance by serial PET Scans | 5 years

SECONDARY OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shyamkishore J Shrivastava, MD, DNB (RT), Principal Investigator — Professor & Head, Radiation Oncology, Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided